CLINICAL TRIAL: NCT02667457
Title: 99mTc-rhAnnexin V-128 Planar and SPECT Imaging of Apoptosis in Asymptomatic Or Previously Symptomatic With TIA Patients With Carotid Atherosclerotic Plaque
Brief Title: 99mTc-rhAnnexin V-128 Imaging for Carotid Atherosclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision based on strategic considerations
Sponsor: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAA-Annexin-04; CAAA113A32201 (Other: Novartis)
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: Carotid Artery Plaque
Keywords: Carotid Stenosis; Carotid Artery Narrowing; Carotid Artery Plaque; Carotid Artery Stenosis; Carotid Artery Ulcerating Plaque; Carotid Ulcer; Common Carotid Artery Stenosis; External Carotid Artery Stenosis; Internal Carotid Artery Stenosis; Plaque, Ulcerating, Carotid Artery; Stenosis, Common Carotid Artery; Stenosis, External Carotid Artery; Ulcerating Plaque, Carotid Artery
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD Participants (Experimental): Participants with asymptomatic or previously symptomatic with TIA only carotid atherosclerotic plaque with evidence of 50% or more carotid stenosis in one or more carotid arteries on carotid ultrasound within 2 years, received a single intravenous bolus of 350 MBq ± 10 % of 99mTc-rhAnnexin V-128 via an intraveneous (IV) catheter in an antecubital vein, followed by a saline flush on screening (Day 0).
  Interventions: Radiation: 99mTc-rhAnnexin V-128
- Healthy Participants (Experimental): Healthy participants with no significant carotid artery disease on carotid ultrasound, received a single intravenous bolus of 350 MBq ± 10 % of 99mTc-rhAnnexin V-128 via an IV catheter in an antecubital vein, followed by a saline flush on screening (Day 0).
  Interventions: Radiation: 99mTc-rhAnnexin V-128

INTERVENTIONS:
Radiation: 99mTc-rhAnnexin V-128

SUMMARY:
This was a single-center, single-dose, study comprising a Proof of Concept (PoC) part and a subsequent Phase II part. The study was being done to assess the ability of the radiotracer 99mTc-rhAnnexin V-128 to image atherosclerotic plaque that might rupture and break off artery walls. This is caused by apoptosis or cell death in the plaque. These ruptured plaques can block blood circulation in the arteries causing a lack of oxygen to the tissues. Atherosclerotic plaques can build up on any artery in the body.

DETAILED DESCRIPTION:
The sponsor decided to terminate the study earlier than planned due to strategic decisions to focus the AAA development portfolio on oncology theragnostics and not based on safety concerns. Novartis acquired Advanced Accelerator Applications SA.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

1. Males and females age 18 years or greater
2. Able and willing to comply with the study procedures
3. Negative pregnancy test for women of childbearing potential at screening and on the day of administration of 99mTc-rhAnnexin V-128.

   For participants with carotid artery disease:
4. Evidence of 50% or more carotid stenosis in one or more carotid arteries on carotid ultrasound within 2 years;
5. Evidence of 50% or more carotid stenosis in the most recent US imaging within 8 weeks prior to 99mTc-rhAnnexin V-128 administration

   For control participants:
6. No significant carotid artery disease on carotid ultrasound;
7. No clinically significant abnormalities in baseline laboratory values.

Exclusion Criteria:

1. Previous carotid stending, endarterectomy or stroke;
2. Diagnosis of vasculitis, dissection, or non-atherosclerotic carotid disease (Ehlers-Danlos, Marfans);
3. Pregnancy or lactation;
4. History of any disease or relevant physical or psychiatric condition or abnormal physical finding which may interfere with the study objectives at the investigator judgment;
5. Know hypersensitivity to the investigational product or any of its components;
6. Claustrophobia or inability to lie still in a supine position;
7. Participation in another clinical trial within 4 weeks before study inclusion, except for patients who have participated or who are currently participating in a study without any study drug administration;
8. Unwillingness to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at single center in Canada.
Pre-assignment Details: A total of 39 participants were screened and enrolled to the study, of which only 36 participants were administered with investigational imaging product. All 36 treated participants completed the study.
Groups:
- Carotid Atherosclerotic Plaque (CAD) Participants: Participants with asymptomatic or previously symptomatic with TIA only carotid atherosclerotic plaque with evidence of 50% or more carotid stenosis in one or more carotid arteries on carotid ultrasound within 2 years, received a single intravenous bolus of 350 MBq ± 10 % of 99mTc-rhAnnexin V-128 via an intraveneous (IV) catheter in an antecubital vein, followed by a saline flush on Day 0.
- Healthy Participants: Healthy participants with no significant carotid artery disease on carotid ultrasound, received a single intravenous bolus of 350 MBq ± 10 % of 99mTc-rhAnnexin V-128 via an IV catheter in an antecubital vein, followed by a saline flush on Day 0.
Period: Overall Study
Arm/Group | Carotid Atherosclerotic Plaque (CAD) Participants | Healthy Participants
Started (All screened/enrolled participants) | 27 | 12
Dosed Participants (All infused enrolled participants were included in Safety Population Set) | 26 | 10
Full Analysis Set Population (FAS) (Dosed participants who completed 99mTc-rhAnnexin V-128 imaging procedure.) | 25 | 10
Completed | 26 | 10
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other Reason | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population Set
Groups:
- CAD Participants: Participants with asymptomatic or previously symptomatic with TIA only carotid atherosclerotic plaque with evidence of 50% or more carotid stenosis in one or more carotid arteries on carotid ultrasound within 2 years, received a single intravenous bolus of 350 MBq ± 10 % of 99mTc-rhAnnexin V-128 via an IV catheter in an antecubital vein, followed by a saline flush on Day 0.
- Total: Total of all reporting groups
Arm/Group | CAD Participants | Healthy Participants | Total
Number analyzed (Participants) | 26 | 10 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (6.6) | 58.4 (12.1) | 67.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 21 | 5 | 26
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 26 | 9 | 35
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Evaluated for Imaging Feasibility
Description: The frequency and severity of abnormal carotid scans was determined in the CAD participants and control groups by review of the number, localization, length and uptake intensity grade of each plaque to define a positive or negative scan at each time point. The feasibility of imaging apoptotic activity in CAD using 99mTc-rhAnnexin V-128 was assessed by the data monitoring committee (visual image review and consensus). The three reviewers of the DMC did an independent visual assessment of the images using a 1 to 4 point grading system: each observer reviewed the images of each patient and scored either 1 or 2 (uptake was less than or equal to blood pool), these images were considered normal; 3 was equivocal and four equalled abnormal. Only descriptive analysis performed.
Time Frame: Day 0
Population: Full Analysis Set population (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | CAD Participants | Healthy Participants
Number analyzed (Participants) | 25 | 10
Participants | 15 | 5

2. Primary Outcome: Percentage of Participants With Prevalence of Abnormal 99mTc-rhAnnexin V-128 SPECT/CT Imaging (Phase II Step)
Description: The prevalence of apoptotic activity was defined as the percentage of participants with "abnormal" Single-Photon Emission Computed Tomography (SPECT) imaging scans (also described as positive scans). The overall result of 99mTc-rhAnnexin V-128 imaging was unique: participants with at least one SPECT imaging as positive result (after 60 min or after 120 min from 99mTc-rhAnnexin V-128 injection) were considered as abnormal, participants with SPECT/CT images as negative were considered as normal. All images were acquired with a dual head SPECT/CT gamma camera with low-energy high-resolution collimators. Only descriptive analysis performed.
Time Frame: At 60 and 120 minutes post injection on Day 0
Population: Full Analysis Set population (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | CAD Participants | Healthy Participants
Number analyzed (Participants) | 25 | 10
Participants
  60 mins after injection: Positive (abnormal) | 8 | 0
  60 mins after injection: Negative (normal) | 16 | 10
  60 mins after injection: Missing | 1 | 0
  120 mins after injection: Positive (abnormal) | 8 | 0
  120 mins after injection: Negative (normal) | 17 | 10
  120 mins after injection: Missing | 0 | 0

3. Secondary Outcome: Left Carotid Uptake Imaging Assessment as Measured by Target to Background Ratio (TBR)
Description: Quantitative analysis of planar images was carried out by placing a region of interest in the carotid areas and over a background area placed in the subclavian regions representing venous and arterial activity (target-to-background). Carotid artery uptake measured as TBR data for right and left carotids at 1 and 2 hours was compared between normal control and carotid artery disease groups.
  Quantitative analysis of the SPECT 1 and 2 hour images was done with regions of interest placed over the arterial target (right carotid, left carotid, ascending aorta, arch and descending aorta) and adjacent vein (internal jugular, SVC or IVS) using transaxial slices. TBR was calculated as arterial max / venous mean (the average of 3 slices centered on the slice with the highest TBR value).
Time Frame: At 60 and 120 minutes post injection on Day 0
Population: Full Analysis Set (FAS). Only participants with Left Carotid Uptake Imaging Assessment included in the analysis.
Measure: Mean (Standard Deviation); unit: Target to Background Ratio (TBR)
Arm/Group | CAD Participants | Healthy Participants
Number analyzed (Participants) | 25 | 10
Target to Background Ratio (TBR)
  60 Minutes: number analyzed (Participants) | 24 | 10
  60 Minutes | 1.171 (0.764) | 0.697 (0.222)
  120 Minutes: number analyzed (Participants) | 24 | 10
  120 Minutes | 1.208 (0.486) | 0.827 (0.205)
Statistical Analysis 1: Comparison: CAD Participants vs Healthy Participants; Timepoint = 60 minutes; Test type: Other; p = 0.0095, t-test, 1 sided — p-value is based on t-test with unequal variances (Satterthwaite) if p-value of F-test for Equality of variances is significant (p<0.05) otherwise p-value is based on t-test with equal variances
Statistical Analysis 2: Comparison: CAD Participants vs Healthy Participants; Timepoint = 120 minutes; Test type: Other; p = 0.0029, t-test, 1 sided — [p-value comment as in outcome 3, analysis 1]

4. Secondary Outcome: Right Carotid Uptake Imaging Assessment as Measured by Target to Background Ratio (TBR)
Description: as for outcome 3
Time Frame: At 60 and 120 minutes post injection on Day 0
Population: Full Analysis Set (FAS). Only participants with Right Carotid Uptake Imaging Assessment included in the analysis.
Measure: Mean (Standard Deviation); unit: Target to Background Ratio (TBR)
Arm/Group | CAD Participants | Healthy Participants
Number analyzed (Participants) | 25 | 10
Target to Background Ratio (TBR)
  60 Minutes: number analyzed (Participants) | 24 | 10
  60 Minutes | 1.252 (0.745) | 0.768 (0.209)
  120 Minutes: number analyzed (Participants) | 24 | 10
  120 Minutes | 1.220 (0.550) | 0.928 (0.217)
Statistical Analysis 1: Comparison: CAD Participants vs Healthy Participants; Timepoint = 60 minutes; Test type: Other; p = 0.0066, t-test, 1 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: CAD Participants vs Healthy Participants; Timepoint = 120 minutes; Test type: Other; p = 0.0334, t-test, 1 sided — [p-value comment as in outcome 3, analysis 1]

5. Secondary Outcome: Ascending Aorta Uptake Imaging Assessment as Measured by Target to Background Ratio (TBR)
Description: as for outcome 3
Time Frame: At 60 and 120 minutes post injection on Day 0
Population: Full Analysis Set (FAS). Only participants with Ascending Aorta Uptake Imaging Assessment included in the analysis.
Measure: Mean (Standard Deviation); unit: Target to Background Ratio (TBR)
Arm/Group | CAD Participants | Healthy Participants
Number analyzed (Participants) | 25 | 10
Target to Background Ratio (TBR)
  60 Minutes: number analyzed (Participants) | 21 | 10
  60 Minutes | 2.054 (0.656) | 1.574 (0.252)
  120 Minutes: number analyzed (Participants) | 20 | 10
  120 Minutes | 1.616 (0.294) | 1.381 (0.190)
Statistical Analysis 1: Comparison: CAD Participants vs Healthy Participants; Timepoint = 60 minutes; Test type: Other; p = 0.0066, t-test, 1 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: CAD Participants vs Healthy Participants; Timepoint = 120 minutes; Test type: Other; p = 0.0301, t-test, 1 sided — [p-value comment as in outcome 3, analysis 1]

6. Secondary Outcome: Descending Aorta Uptake Imaging Assessment as Measured by Target to Background Ratio (TBR)
Description: as for outcome 3
Time Frame: At 60 and 120 minutes post injection on Day 0
Population: Full Analysis Set (FAS). Only participants with Descending Aorta Uptake Imaging Assessment included in the analysis.
Measure: Mean (Standard Deviation); unit: Target to Background Ratio (TBR)
Arm/Group | CAD Participants | Healthy Participants
Number analyzed (Participants) | 25 | 10
Target to Background Ratio (TBR)
  60 Minutes: number analyzed (Participants) | 22 | 10
  60 Minutes | 2.159 (0.865) | 1.590 (0.164)
  120 Minutes: number analyzed (Participants) | 21 | 10
  120 Minutes | 1.520 (0.245) | 1.341 (0.131)
Statistical Analysis 1: Comparison: CAD Participants vs Healthy Participants; Timepoint = 60 minutes; Test type: Other; p = 0.0066, t-test, 1 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: CAD Participants vs Healthy Participants; Timepoint = 120 minutes; Test type: Other; p = 0.0387, t-test, 1 sided — [p-value comment as in outcome 3, analysis 1]

7. Secondary Outcome: Aortic Arch Uptake Correlation Imaging Assessment as Measured by Target to Background Ratio (TBR)
Description: as for outcome 3
Time Frame: At 60 and 120 minutes post injection on Day 0
Population: Full Analysis Set (FAS). Only participants with Aortic Arch Uptake Correlation Imaging Assessment included in the analysis.
Measure: Mean (Standard Deviation); unit: Target to Background Ratio (TBR)
Groups:
- CAD Participants: Participants with asymptomatic carotid atherosclerotic plaque or previously symptomatic with TIA only with evidence of 50% or more carotid stenosis in one or more carotid arteries on carotid ultrasound within 2 years, received a single intravenous bolus of 350 MBq ± 10 % of 99mTc-rhAnnexin V-128 via an IV catheter in an antecubital vein, followed by a saline flush on Day 0.
Arm/Group | CAD Participants | Healthy Participants
Number analyzed (Participants) | 25 | 10
Target to Background Ratio (TBR)
  60 Minutes: number analyzed (Participants) | 22 | 10
  60 Minutes | 1.986 (0.679) | 1.606 (0.279)
  120 Minutes: number analyzed (Participants) | 21 | 10
  120 Minutes | 1.628 (0.380) | 1.294 (0.174)
Statistical Analysis 1: Comparison: CAD Participants vs Healthy Participants; Timepoint = 60 minutes; Test type: Other; p = 0.0359, t-test, 1 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: CAD Participants vs Healthy Participants; Timepoint = 120 minutes; Test type: Other; p = 0.0022, t-test, 1 sided — [p-value comment as in outcome 3, analysis 1]

8. Secondary Outcome: Left Carotid Uptake Imaging Assessment as Measure by Target to Background Ratio (TBR) by Ultrasound Grade of Plaque Echolucency/Echogenicity
Description: B-mode and color Doppler ultrasound studies were acquired of both carotid arteries and performed with an ultrasound scanner equipped with a 5- to 7-MHz transducer. Plaque morphology, as echogenicity, defined as reflectance of the emitted ultrasound signal, were assessed and graded from 1 to 4 as echolucent, predominantly echolucent, predominantly echogenic, or echogenic. The vessel lumen was used as the reference structure for defining echolucency, and the bright echo zone produced by the media-adventitia interface in the far wall was used as the reference structure for defining echogenicity. Uptake was reported as the ratio of the uptake in the region of interest (target) to the uptake in the blood pool (background). Only descriptive analysis performed.
Time Frame: At 60 and 120 minutes post injection on Day 0
Population: Full Analysis Set (FAS). Only participants with left carotid with stenosis >=50% are taken into account.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | CAD Participants
Number analyzed (Participants) | 25
Ratio
  Echolucent: 60 Minutes: number analyzed (Participants) | 0
  Echolucent: 120 Minutes: number analyzed (Participants) | 0
  Predominantly echolucent: 60 Minutes: number analyzed (Participants) | 3
  Predominantly echolucent: 60 Minutes | 1.490 (0.756)
  Predominantly echolucent: 120 Minutes: number analyzed (Participants) | 3
  Predominantly echolucent: 120 Minutes | 1.014 (0.309)
  Predominantly echogenic: 60 Minutes: number analyzed (Participants) | 7
  Predominantly echogenic: 60 Minutes | 0.945 (0.287)
  Predominantly echogenic: 120 Minutes: number analyzed (Participants) | 7
  Predominantly echogenic: 120 Minutes | 1.096 (0.186)
  Echogenic: 60 Minutes: number analyzed (Participants) | 6
  Echogenic: 60 Minutes | 0.950 (0.245)
  Echogenic: 120 Minutes: number analyzed (Participants) | 6
  Echogenic: 120 Minutes | 1.387 (0.496)

9. Secondary Outcome: Right Carotid Uptake Imaging Assessment as Measure by Target to Background Ratio (TBR) by Ultrasound Grade of Plaque Echolucency/Echogenicity
Description: as for outcome 8
Time Frame: At 60 and 120 minutes post injection on Day 0
Population: Full Analysis Set (FAS). Only participants with right carotid with stenosis >=50% are taken into account.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | CAD Participants
Number analyzed (Participants) | 25
Ratio
  Echolucent: 60 Minutes: number analyzed (Participants) | 1
  Echolucent: 60 Minutes | 0.619 (0.000)
  Echolucent: 120 Minutes: number analyzed (Participants) | 1
  Echolucent: 120 Minutes | 0.820 (0.000)
  Predominantly echolucent: 60 Minutes: number analyzed (Participants) | 7
  Predominantly echolucent: 60 Minutes | 0.955 (0.192)
  Predominantly echolucent: 120 Minutes: number analyzed (Participants) | 7
  Predominantly echolucent: 120 Minutes | 1.126 (0.311)
  Predominantly echogenic: 60 Minutes: number analyzed (Participants) | 8
  Predominantly echogenic: 60 Minutes | 1.593 (1.174)
  Predominantly echogenic: 120 Minutes: number analyzed (Participants) | 8
  Predominantly echogenic: 120 Minutes | 1.294 (0.851)
  Echogenic: 60 Minutes: number analyzed (Participants) | 4
  Echogenic: 60 Minutes | 1.180 (0.206)
  Echogenic: 120 Minutes: number analyzed (Participants) | 4
  Echogenic: 120 Minutes | 1.149 (0.438)

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious AEs and Death
Description: An AE is defined as any untoward medical occurrence in a participant and which does not necessarily have a causal relationship with the investigational product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease, temporally associated with the use of an investigational product, whether or not causally related to the investigational product. Treatment emergent adverse events that emerge after the 99mTc-rhAnnexin V-128 injection and up to 30 days after the injection that were absent before it or worsen relative to the pre-treatment state. A serious AE is defined as any untoward medical occurrence that at any dose results in death; is life-threatening; results in persistent or significant disability or incapacity; results in congenital anomaly or birth defect; or requires inpatient hospitalization or prolongation of hospitalization. Only descriptive analysis performed.
Time Frame: From Day 0 post injection up to Day 30
Population: Safety Population Set
Measure: Count of Participants; unit: Participants
Arm/Group | CAD Participants | Healthy Participants
Number analyzed (Participants) | 26 | 10
Participants
  Treatment Emergent Adverse Events (TEAEs) | 7 | 0
  Treatment Emergent Adverse Drug Reactions | 2 | 0
  Treatment Emergent Serious Adverse Events (TESAEs) | 1 | 0
  Treatment Emergent Serious Adverse Drug Reactions | 0 | 0
  TEAEs leading to Withdrawal | 0 | 0
  TEAEs leading to Deaths | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Values
Description: Laboratory data was analysed with respect to the normal ranges of values provided by the local laboratory and with respect to levels of change and significance in these values. The evaluation of the "Clinically Significant Abnormal Laboratory Values" was at the discretion of the Principal Investigator and noted as such in patient files, where necessary. Participants with abnormal laboratory values were analyzed based on clinical relevance. Only descriptive analysis performed.
Time Frame: From Day 0 post injection up to Day 30
Population: Safety Population Set. Only participants with abnormal laboratory values are taken into account.
Measure: Count of Participants; unit: Participants
Arm/Group | CAD Participants | Healthy Participants
Number analyzed (Participants) | 26 | 10
Participants
  Blood Chemistry: Abnormal non clinical relevant | 26 | 10
  Blood Chemistry: Abnormal clinically relevant | 0 | 0
  Hematology: number analyzed (Participants) | 15 | 4
  Hematology: Abnormal non clinical relevant | 15 | 4
  Hematology: Abnormal clinically relevant | 0 | 0
  Urinalysis: number analyzed (Participants) | 10 | 4
  Urinalysis: Abnormal non clinical relevant | 10 | 4
  Urinalysis: Abnormal clinically relevant | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 0 up to Day 30
Description: Analysis was performed in the safety population defined as all participants who received the administration of 99mTc-rhAnnexin V-128.
Groups:
- CAD Participants: Participants with asymptomatic carotid atherosclerotic plaque or previously symptomatic with TIA only with evidence of 50% or more carotid stenosis in one or more carotid arteries on carotid ultrasound within 2 years, received a single intravenous bolus of 350 MBq ± 10 % of 99mTc-rhAnnexin V-128 via an IV catheter in an antecubital vein, followed by a saline flush on screening (Day 0).
Arm/Group | CAD Participants | Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/10
Other Adverse Events (participants affected / at risk) | 7/26 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAD Participants (N=26) | Healthy Participants (N=10)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAD Participants (N=26) | Healthy Participants (N=10)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Claustrophobia (Psychiatric disorders) | 1 (1) | 0 (0)
Sinus headache (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was prematurely terminated on 19-Mar-2019 due to strategic decisions to focus the AAA development portfolio on oncology theragnostics, and not based on any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT02667457/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT02667457/SAP_001.pdf